CLINICAL TRIAL: NCT01444664
Title: Aneurysm Wall Histology and Correlation With Cerebrospinal Fluid and Blood Plasma Registry
Brief Title: Aneurysm Wall Histology Registry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Albany Medical College (Other); Northwestern University (Other); Stony Brook University (Other); Royal University Hospital Foundation (Other); Indiana University (Other); Providence Health & Services (Other); University of Illinois at Chicago (Other); Vanderbilt University (Other); Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20137
Record Dates: First submitted 2011-08-30; First posted 2011-10-03 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2015-04

CONDITIONS: Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aneurysm (Experimental)
  Interventions: Procedure: Surgical Clipping of Aneurysm

INTERVENTIONS:
Procedure: Surgical Clipping of Aneurysm — Surgical clipping of intracranial aneurysm

SUMMARY:
The purpose of this prospective registry is to determine if patients harboring intracranial aneurysms have any predictive markers between aneurysm wall tissue, cerebrospinal fluid and blood plasma.

DETAILED DESCRIPTION:
To design a registry to evaluate the wall of intracranial aneurysms during open surgical clipping by direct photographic appearance, wall biopsy samples, CSF and blood plasma fluid collection (Interleukins; IL-8/ Matrix Metalloproteinase; MMP-9) for complete evaluation and comparison.

The focus of the registry will be to determine the presence of aneurysmal wall defects, mural clot, atherosclerotic and atheroma, wall permeability and delamination. These findings will then be correlated to the collected CSF and blood values to determine if there is any direct features of the aneurysm wall that would predict any of the reported post embolic syndromes. The collected data can also be correlated to the peroperative imaging, (MRI, CT and Angiogram).

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years but < 80 years of age
* Patient with an unruptured Intracranial aneurysm 8mm or larger
* Patient that surgical exposure and clipping will be the primary treatment option

Exclusion Criteria:

* Any patient that has a ruptured intracranial aneurysm
* Any Pediatric patients
* Any patient presenting with any pre-treatment intracranial lesions

  * Vascular malformations
  * Hemorrhage
  * Normal Pressure Hydrocephalus
  * Obstructive Hydrocephalus
  * White matter disease
  * Tumors
  * Trauma
  * Other vascular type lesions
* Any meningitis type symptoms
* Medical or surgical co-morbidities such that the patient's life expectancy is less than 1 year
* Inability to obtain consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Histological Change | an average of 1 day after aneurysm treatment an analysis of the histological sample, CSF sample, and plasma samples will occur
  To determine the relative and absolute differences in histological changes as seen in the tissue samples comparing this to the CSF and blood plasma samples. To also determine if there is any gene expressions that can be utilized as predictive markers in this cohort of patients.

SECONDARY OUTCOMES:
Treatment related morbidity and mortality | up to approximately 1 year post treatment
  Secondary analyses will be performed to compare treatment related morbidity and mortality,
Clinical Outcome | approximately clinical outcome at 6 months after surgical clipping at routine follow up visit and approximately 12 months after clipping at routine follow up visit if indicated
  clinical outcome at approximately 6 months after surgical clipping at routine follow up visit and approximately 12 months after clipping at routine follow up visit if indicated
Bleeding Rate | post treatment during approximate follow up periods 6mo and 12mo clinical follow up
  bleeding rate post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Woo, Principal Investigator — SUNY - Stonybrook; Arthur Adam, MD, Principal Investigator — Baptist Hospital; Mike Kelly, Principal Investigator — Royal University Hospital Foundation
Locations (10):
- United States (9):
  - Northwestern University, Chicago, Illinois
  - University Of Illinois, Chicago, Illinois
  - Goodman Campbell, Indianapolis, Indiana
  - Albany Medical Center, Albany, New York
  - SUNY - Stonybrook University Medical Center, Stony Brook, New York
  - Providence Health, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Healthcare - Memphis, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
- Royal University Hospital, Saskatoon, Ontario, Canada

REFERENCES:
- [Background] Weir B. Unruptured intracranial aneurysms: a review. J Neurosurg. 2002 Jan;96(1):3-42. doi: 10.3171/jns.2002.96.1.0003. PMID 11794601
- [Background] Ronkainen A, Hernesniemi J. Subarachnoid haemorrhage of unknown aetiology. Acta Neurochir (Wien). 1992;119(1-4):29-34. doi: 10.1007/BF01541778. PMID 1481749
- [Background] STEHBENS WE. ANEURYSMS AND ANATOMICAL VARIATION OF CEREBRAL ARTERIES. Arch Pathol. 1963 Jan;75:45-64. No abstract available. PMID 14087271
- [Background] Brisman JL, Song JK, Newell DW. Cerebral aneurysms. N Engl J Med. 2006 Aug 31;355(9):928-39. doi: 10.1056/NEJMra052760. No abstract available. PMID 16943405
- [Background] Juvela S, Hillbom M, Numminen H, Koskinen P. Cigarette smoking and alcohol consumption as risk factors for aneurysmal subarachnoid hemorrhage. Stroke. 1993 May;24(5):639-46. doi: 10.1161/01.str.24.5.639. PMID 8488517
- [Background] Juvela S. Prehemorrhage risk factors for fatal intracranial aneurysm rupture. Stroke. 2003 Aug;34(8):1852-7. doi: 10.1161/01.STR.0000080380.56799.DD. Epub 2003 Jun 26. PMID 12829865
- [Background] Sahs AL. Observations on the pathology of saccular aneurysms. J Neurosurg. 1966 Apr;24(4):792-806. doi: 10.3171/jns.1966.24.4.0792. No abstract available. PMID 5934137
- [Background] Scanarini M, Mingrino S, Giordano R, Baroni A. Histological and ultrastructural study of intracranial saccular aneurysmal wall. Acta Neurochir (Wien). 1978;43(3-4):171-82. doi: 10.1007/BF01587953. PMID 707175
- [Background] Krex D, Schackert HK, Schackert G. Genesis of cerebral aneurysms--an update. Acta Neurochir (Wien). 2001;143(5):429-48; discussion 448-9. doi: 10.1007/s007010170072. PMID 11482693
- [Background] Kataoka K, Taneda M, Asai T, Kinoshita A, Ito M, Kuroda R. Structural fragility and inflammatory response of ruptured cerebral aneurysms. A comparative study between ruptured and unruptured cerebral aneurysms. Stroke. 1999 Jul;30(7):1396-401. doi: 10.1161/01.str.30.7.1396. PMID 10390313
- [Background] Chyatte D, Bruno G, Desai S, Todor DR. Inflammation and intracranial aneurysms. Neurosurgery. 1999 Nov;45(5):1137-46; discussion 1146-7. doi: 10.1097/00006123-199911000-00024. PMID 10549930
- [Background] Bruno G, Todor R, Lewis I, Chyatte D. Vascular extracellular matrix remodeling in cerebral aneurysms. J Neurosurg. 1998 Sep;89(3):431-40. doi: 10.3171/jns.1998.89.3.0431. PMID 9724118
- [Background] Nakajima N, Nagahiro S, Sano T, Satomi J, Satoh K. Phenotypic modulation of smooth muscle cells in human cerebral aneurysmal walls. Acta Neuropathol. 2000 Nov;100(5):475-80. doi: 10.1007/s004010000220. PMID 11045669
- [Background] Kosierkiewicz TA, Factor SM, Dickson DW. Immunocytochemical studies of atherosclerotic lesions of cerebral berry aneurysms. J Neuropathol Exp Neurol. 1994 Jul;53(4):399-406. doi: 10.1097/00005072-199407000-00012. PMID 8021714
- [Background] Aydin F. Do human intracranial arteries lack vasa vasorum? A comparative immunohistochemical study of intracranial and systemic arteries. Acta Neuropathol. 1998 Jul;96(1):22-8. doi: 10.1007/s004010050856. PMID 9678510
- [Background] Ushikoshi S, Kikuchi Y, Houkin K, Miyasaka K, Abe H. Aggravation of brainstem symptoms caused by a large superior cerebellar artery aneurysm after embolization by Guglielmi detachable coils--case report. Neurol Med Chir (Tokyo). 1999 Jul;39(7):524-9. doi: 10.2176/nmc.39.524. PMID 10437381
- [Background] Meyers PM, Lavine SD, Fitzsimmons BF, Commichau C, Parra A, Mayer SA, Solomon RA, Connolly ES Jr. Chemical meningitis after cerebral aneurysm treatment using two second-generation aneurysm coils: report of two cases. Neurosurgery. 2004 Nov;55(5):1222. doi: 10.1227/01.neu.0000140987.71791.df. PMID 15791738
- [Background] Berenstein A, Song JK, Niimi Y, Namba K, Heran NS, Brisman JL, Nahoum MC, Madrid M, Langer DJ, Kupersmith MJ. Treatment of cerebral aneurysms with hydrogel-coated platinum coils (HydroCoil): early single-center experience. AJNR Am J Neuroradiol. 2006 Oct;27(9):1834-40. PMID 17032853
- [Background] Bendszus M, Solymosi L. Cerecyte coils in the treatment of intracranial aneurysms: a preliminary clinical study. AJNR Am J Neuroradiol. 2006 Nov-Dec;27(10):2053-7. PMID 17110665
- [Background] Deshaies EM, Adamo MA, Boulos AS. A prospective single-center analysis of the safety and efficacy of the hydrocoil embolization system for the treatment of intracranial aneurysms. J Neurosurg. 2007 Feb;106(2):226-33. doi: 10.3171/jns.2007.106.2.226. PMID 17410704
- [Background] Im SH, Han MH, Kwon BJ, Jung C, Kim JE, Han DH. Aseptic meningitis after embolization of cerebral aneurysms using hydrogel-coated coils: report of three cases. AJNR Am J Neuroradiol. 2007 Mar;28(3):511-2. PMID 17353325
- [Background] Stracke CP, Krings T, Moller-Hartmann W, Mahdavi A, Klug N. Severe inflammatory reaction of the optic system after endovascular treatment of a supraophthalmic aneurysm with bioactive coils. AJNR Am J Neuroradiol. 2007 Aug;28(7):1401-2. doi: 10.3174/ajnr.A0550. PMID 17698551
- [Background] Schmidt GW, Oster SF, Golnik KC, Tumialan LM, Biousse V, Turbin R, Prestigiacomo CJ, Miller NR. Isolated progressive visual loss after coiling of paraclinoid aneurysms. AJNR Am J Neuroradiol. 2007 Nov-Dec;28(10):1882-9. doi: 10.3174/ajnr.A0690. PMID 17998416
- [Background] Kang HS, Han MH, Lee TH, Shin YS, Roh HG, Kwon OK, Kwon BJ, Kim SY, Kim SH, Byun HS. Embolization of intracranial aneurysms with hydrogel-coated coils: result of a Korean multicenter trial. Neurosurgery. 2007 Jul;61(1):51-8; discussion 58-9. doi: 10.1227/01.neu.0000279723.67779.f0. PMID 17621018
- [Background] Pickett GE, Laitt RD, Herwadkar A, Hughes DG. Visual pathway compromise after hydrocoil treatment of large ophthalmic aneurysms. Neurosurgery. 2007 Oct;61(4):E873-4; discussion E874. doi: 10.1227/01.NEU.0000298918.55119.7C. PMID 17986922
- [Background] Horie N, Kitagawa N, Morikawa M, Tsutsumi K, Kaminogo M, Nagata I. Progressive perianeurysmal edema induced after endovascular coil embolization. Report of three cases and review of the literature. J Neurosurg. 2007 May;106(5):916-20. doi: 10.3171/jns.2007.106.5.916. PMID 17542541
- [Background] Marchan EM, Sekula RF Jr, Ku A, Williams R, O'Neill BR, Wilberger JE, Quigley MR. Hydrogel coil-related delayed hydrocephalus in patients with unruptured aneurysms. J Neurosurg. 2008 Aug;109(2):186-90. doi: 10.3171/JNS/2008/109/8/0186. PMID 18671628
- [Background] Fanning NF, Willinsky RA, ter Brugge KG. Wall enhancement, edema, and hydrocephalus after endovascular coil occlusion of intradural cerebral aneurysms. J Neurosurg. 2008 Jun;108(6):1074-86. doi: 10.3171/JNS/2008/108/6/1074. PMID 18518706
- [Background] White JB, Cloft HJ, Kallmes DF. But did you use HydroCoil? Perianeurysmal edema and hydrocephalus with bare platinum coils. AJNR Am J Neuroradiol. 2008 Feb;29(2):299-300. doi: 10.3174/ajnr.A0877. Epub 2007 Nov 16. PMID 18024573
- [Background] Marden FA, Putman CM. Perianeurysm edema with second-generation bioactive coils. Surg Neurol. 2008 Jun;69(6):627-32; discussion 632. doi: 10.1016/j.surneu.2007.01.069. Epub 2007 Oct 31. PMID 17976696
- [Background] Turner RD, Byrne JV, Kelly ME, Mitsos AP, Gonugunta V, Lalloo S, Rasmussen PA, Fiorella D. Delayed visual deficits and monocular blindness after endovascular treatment of large and giant paraophthalmic aneurysms. Neurosurgery. 2008 Sep;63(3):469-74; discussion 474-5. doi: 10.1227/01.NEU.0000324730.37144.4B. PMID 18812958
- [Background] Im SH, Han MH, Kwon OK, Kwon BJ, Kim SH, Kim JE, Oh CW. Endovascular coil embolization of 435 small asymptomatic unruptured intracranial aneurysms: procedural morbidity and patient outcome. AJNR Am J Neuroradiol. 2009 Jan;30(1):79-84. doi: 10.3174/ajnr.A1290. Epub 2008 Sep 3. PMID 18768715
- [Background] Killer M, Baltsavias G, Huemer M, Richling B. Visual worsening after incomplete coiling of a small asymptomatic aneurysm: case report and review of the literature. Minim Invasive Neurosurg. 2009 Feb;52(1):39-43. doi: 10.1055/s-0028-1104565. Epub 2009 Feb 26. PMID 19247904
- [Background] Nishino K, Ito Y, Hasegawa H, Shimbo J, Kikuchi B, Fujii Y. Development of cranial nerve palsy shortly after endosaccular embolization for asymptomatic cerebral aneurysm: report of two cases and literature review. Acta Neurochir (Wien). 2009 Apr;151(4):379-83. doi: 10.1007/s00701-009-0234-4. Epub 2009 Mar 5. PMID 19262981
- [Background] Hara A, Yoshimi N, Mori H. Evidence for apoptosis in human intracranial aneurysms. Neurol Res. 1998 Mar;20(2):127-30. doi: 10.1080/01616412.1998.11740494. PMID 9522347